CLINICAL TRIAL: NCT06589895
Title: Correlation Between RISANKIZUMAB's Trough Levels, Clinical and Biological Remission in Moderate to Severe Crohn's Disease: a Retrospective Multicentric Study
Acronym: RISE-CD
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2024/LS-01
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to determine if, as with other therapeutics such as anti-TNF, trough levels of Risankizumab are correlated with clinical and biological remission in patients with moderate to severe Crohn's disease. As part of their regular biological surveillance, trough levels of Risankizumab were mesured and clinical and biological data were collected to determine if biological and clinical remission criteria were met.

DETAILED DESCRIPTION:
The treatment of chronic inflammatory bowel disease has undergone a number of therapeutic revolutions in recent years, with the emergence of new biotherapies. These include RISANKIZUMAB, an anti-IL23 p19, whose ADVANCE , MOTIVATE and FORTIFY studies have demonstrated its efficacy in the induction and maintenance phases of Crohn's disease. Reimbursement in France for this indication is expected in the final quarter of 2024.

While for first-line molecules such as anti-TNF alpha, the relationship between serum levels and clinical remission is accepted and allows to guide the therapeutic strategy for patients, it has yet to be demonstrated for new molecules of interest.

We enrolled patients with moderate to severe Crohn's disease on Risankizumab in four centers. Trough levels of Risankizumab were mesured as a part of their regular medical surveillance routine. For each consultation, biological and clinical data were collected to determine wether patients were in remission (according to our primary outcome) or not. Data were collected up to 18 months since the introduction of Risankizumab.

The objectives of this study were also to identify factors of primary or secondary failure of treatment, to determine clinical reponse rate, to evaluate tolerance and persistence of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patients with moderate to severe Crohn's disease
* Failure of at least one immunosuppressant and one anti-TNF alpha agent
* Patients on Risankizumab
* No opposition to study participation

Exclusion Criteria:

* Age < 18 years
* UC
* Unclassified colitis
* Risankizumab prescribed to prevent post-operative relapse
* Any contraindication to Risankizumab
* Refusal to participate in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to severe Crohn's disease on Risankizumab
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Clinical and biological remission without corticosteroids 12 months after introduction of RISANKIZUMAB treatment. | 12 months
  Defined by Harvey-Bradshaw score (HBI < 4) and CRP < 5 mg/L and/or calprotectin < 250 µg/g.

SECONDARY OUTCOMES:
Predictive factors for primary or secondary treatment failure | 18 months
Risk factors for immunisation | 18 months
Risk factors for sub-therapeutics trough levels | 18 months
Clinical response rates | 6 months, 12 months and 18 months
Clinical and biological remission rates | 6 months and 18 months
Drug discontinuation rates | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Nîmes, Nîmes, Gard, France

IPD SHARING:
Plan to Share IPD: No